CLINICAL TRIAL: NCT03617302
Title: Effects of Inorganic Nitrate Supplementation on Cerebrovascular Aging and Arterial Stiffness Study
Brief Title: Inorganic Nitrate Supplementation on Cerebrovascular Aging and Arterial Stiffness Study
Acronym: INCA
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gary L. Pierce (Other)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor-Investigator, Gary L. Pierce, Principle Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 201805720
Record Dates: First submitted 2018-07-30; First posted 2018-08-06 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Aging; Arterial Stiffness; Endothelial Dysfunction; Hypertension; Cognitive Decline
Keywords: Carotid artery stiffness; Cerebrovascular function; Cerebral blood flow; Pulsatility; Beetroot juice; Dietary Inorganic Nitrate Supplementation; Cerebral Small Vessel Disease; Cerebrovascular Reserve; Neurovascular Coupling
MeSH Terms: conditions — Hypertension; Cognitive Dysfunction; Cerebral Small Vessel Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Beetroot juice (Experimental): 10-grams of nitrate-containing beetroot concentrate diluted in 120-180 milliliters of water.
  Interventions: Drug: Experimental: Nitrate-containing
- Placebo Beetroot juice (Placebo Comparator): 10 grams of nitrate-depleted beetroot concentrate balanced for anti-oxidant content diluted in 120-180 milliliters of water.
  Interventions: Drug: Placebo: Nitrate-depleted

INTERVENTIONS:
Drug: Experimental: Nitrate-containing — Experimental
  Arms: Beetroot juice
Drug: Placebo: Nitrate-depleted — Placebo
  Arms: Placebo Beetroot juice

SUMMARY:
This study investigates the effect of dietary inorganic nitrate supplementation on 1) large elastic artery stiffness and hemodynamics and 2) cerebrovascular function in middle-aged and older adults. Participants will be randomized to consume either nitrate-containing or nitrate-depleted beetroot juice.

DETAILED DESCRIPTION:
Reduced nitric oxide bioavailability with aging contributes in part to increased large central artery stiffness and cerebrovascular dysfunction. Large central artery stiffness is a risk factor for cognitive decline mediated in part by the development of cerebrovascular dysfunction. This study will investigate the degree to which improving nitric oxide bioavailability using dietary inorganic nitrate supplementation improves cerebrovascular function through reductions in large central artery stiffness in middle-aged and older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-79 years
* Cognitively healthy, having mild cognitive impairment
* Able to undergo cardiovascular testing procedures including fasting overnight and holding selected morning medication doses.
* Ability to understand and willingness to sign a written informed consent document.
* Ability to lie comfortably for up to 90 minutes
* Women only: Post-menopausal

Exclusion Criteria:

* Current or history of cardiovascular disease disease (heart attack, stroke, heart failure, cardiomyopathy or peripheral artery disease, heart angioplasty/stent or bypass surgery, valve replacement, carotid endarterectomy, heart transplant.
* Medical history of stroke or other neurological disorder or systemic illness that could potentially affect cognition or brain function (outside of a diagnosis of Mild Cognitive impairment, Alzheimer's Disease) or could affect their safety or comfort while undergoing the imaging or cardiovascular studies.
* Subjects with evidence of cardiovascular disease at baseline or during the exercise test (evidence of myocardial infarction, abnormal cardiac arrhythmia, myocardial ischemia, conduction delays, >1mm S-T segment depression or elevation; >3 beat ventricular tachycardia; atrial fibrillation) will be excluded from the study.
* Wilson's disease, hemochromatosis
* Individuals taking clonidine or other short-acting beta blocker
* Resting blood pressure > 200/ 110 mmHg or systolic <90 mmHg
* Medical history of chronic major psychiatric or current diagnosis of major psychiatric disease (other than dementia).
* Systemic illness or neurological disorder potentially affecting cognition or cerebral blood flow other than mild cognitive impairment
* Unable to provide informed consent due to cognitive impairment
* Currently taking medications that may affect cerebral blood flow (e.g. papaverine, indomethacin, acetazolamide, etc) or efficacy of beetroot juice (proton pump inhibitors)
* Current clinically abnormal thyroid function not adequately regulated by thyroid hormone supplementation or medication.
* Allergic to beets
* Current tobacco user or history of tobacco use within the past 3 months (cigarettes, cigars, chewing tobacco, hookah, electronic cigarettes) or living with someone who smokes/has smoked in the past 3 months.
* Current diagnosis of insulin-dependent diabetes (Type I or insulin dependent Type II)
* Current diagnosis of chronic obstructive lung disease, cystic fibrosis, emphysema, chronic bronchitis
* History of renal failure, dialysis or kidney transplant
* Current diagnosis or history of liver disease or HIV/AIDS, or cancer (other than non-melanoma skin cancers).
* Current diagnosis or history of rheumatoid arthritis, systemic lupus erythematosus, Wegener's granulomatosis
* Vulnerable populations (prisoners, etc) will not be eligible.
* Unwillingness to wash out from a vitamin or dietary supplement regime prior to enrollment and maintain throughout the duration of the study.
* Inability to comply with experimental instructions.
* Uncontrolled intercurrent illness that would limit compliance with study requirements per investigator.
* Inability to fast or hold morning medications doses until after testing is complete.
* Hormone replacement use within the past 6 months
* Currently enrolled in another study using an study medication, supplement, device or intervention.

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Acute change in carotid artery stiffness | 2-hours
  Common carotid artery stiffness measured by ultrasonography and applanation tonometry.
Acute change in cerebral blood flow | 2-hours
  Large cerebral artery blood flow will be measured using 4-Dimensional (4D) phase contrast vastly undersampled isotropic projection imaging (pcVIPR) magnetic resonance imaging (MRI).

CONTACTS AND LOCATIONS:
Overall Officials: Gary Pierce, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No